CLINICAL TRIAL: NCT00858611
Title: VRC 307: A D/B Randomized Ph. I Study of Safety/Immunogenicity of a Prime-Boost Schedule of an Investigational DNA Influenza Vaccine, Followed by the Seasonal Influenza Trivalent Inactivated Vaccine (TIV), Compared to TIV Alone in Healthy Adults
Brief Title: VRC 307: A Double-Blind, Randomized Phase I Study of the Safety and Immunogenicity of a Prime-Boost Schedule of the Investigational DNA Trivalent Influenza Vaccine, VRC-FLUDNA047-00-VP, Followed by the 2008/2009 Seasonal Influenza Trivalent Inactivat...
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: RCHSPB
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 090090; 09-I-0090
Record Dates: First submitted 2009-03-07; First posted 2009-03-10 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-06-21

CONDITIONS: Influenza, Human
Keywords: Influenza; Healthy; Immunity; Preventive; Flu; Healthy Volunteer; HV
MeSH Terms: conditions — Influenza, Human | interventions — FluLaval

INTERVENTIONS:
Drug: VRC-FLUDNA047-00-VP
Drug: Flulaval (Registered) Seasonal Influenza Vaccine

SUMMARY:
Objectives:

* To evaluate the safety and tolerability of a prime-boost study regimen that includes the recombinant DNA vaccine followed by licensed 2008/2009 FluLaval(Registered Trademark) in adults ages 18-50 years and adults ages 51-70 years as compared with control groups that receive the licensed vaccine only.
* To evaluate whether the study participants in each age group receiving a prime-boost schedule have a greater frequency of H1 or H3 neutralizing antibodies compared with those of the same age group who received only the 2008/2009 trivalent influenza vaccine.
* To evaluate differences in antibody or T cell responses (quantity, quality, or durability) between the two groups.

Eligibility:

* Participants ages 18 to 70 years of age who are available for clinic follow-up through Week 24 and who have no previously undiagnosed clinically significant chronic diseases. Participants will provide blood samples for further testing to determine eligibility. Females must not be or become pregnant during the study.
* Volunteers who have been immunized with the current season FDA-approved influenza vaccine (2008-2009), or who are being treated for tuberculosis may not participate.

Design:

* The study lasts for 24 weeks.
* Week 0: The first day of Week 0 (i.e., Day 0) is defined as the day of enrollment and first injection. Specific eligibility is reviewed. Participants will receive an injection of either the DNA vaccine VRC-FLUDNA047-00-VP (at 4 mg dosage) or a placebo.
* Week 4: All study participants will receive an injection of the trivalent seasonal influenza vaccine, according to the manufacturer's package insert directions.
* Participants will be given 7-day diary cards on which to record temperature and symptoms (e.g., muscle aches, headache, chills, nausea) and injection site reactions (e.g., pain, tenderness). Participants may also enter this information via the Internet. Presence of symptoms may require additional visits to the clinic.
* Participants will return to the clinic 2 weeks after each injection for the following procedures:
* Blood draws for further tests to determine the immune system's response to the vaccine(s) Clinical evaluations: vital signs and weight, examinations of the lymph nodes, and targeted physical exam on any visit if indicated by interim complaints or laboratory findings.

DETAILED DESCRIPTION:
Study Design:

This is a Phase I, randomized study in healthy younger (18-50 years) and older (51-70 years) adults. For each age group, the study will evaluate the safety, tolerability, and immunogenicity of a prime-boost vaccination regimen against the seasonal influenza virus with an investigational plasmid DNA vaccine as a prime followed 4 weeks later by the seasonal influenza trivalent inactivated vaccine (TIV) boost as compared to the seasonal TIV alone. Equal numbers of healthy adults in each age group will receive the DNA vaccine as the first injection or a control injection with phosphate buffered saline (PBS) as the first injection. The hypothesis is that the DNA vaccine will be safe for human administration and that the prime-boost schedule will elicit a higher titer antibody response than the seasonal TIV alone. The primary objectives are to evaluate the safety and tolerability and induced antibody titer of the investigational prime-boost regimen, at a dose of 4 mg for the DNA vaccine and 45 micrograms ((Micro)g) for the seasonal TIV vaccine. Secondary and exploratory objectives are related to the humoral and cellular immune responses.

Product Description:

The inactivated seasonal influenza vaccine is the trivalent subunit virion vaccine for the 2008-2009 season. Each dose is composed of 45 (Micro)g hemagglutinin (HA) in 0.5 mL; with the recommended ratio of 15 (Micro)g HA of each of the following 3 strains: A/Brisbane/59/2007-like (H1N1); A/Brisbane/10/2007-like (H3N2), A/Uruguay/716/2007, and B/Florida/4/2006-like. The VRC-FLUDNA047-00-VP vaccine was developed and manufactured by VRC, NIAID and is composed of 3 closed-circular DNA plasmids, each with a CMV/R promoter that encode for 2008-2009 strains of the H1, H3 and B proteins. DNA vaccine vials will be supplied at 4 mg/mL and each dose will be 1 mL. The placebo for the DNA vaccine is PBS. Vaccination will be administered intramuscularly (IM) in the deltoid muscle using needle and syringe for the seasonal influenza vaccine and the Biojector(Registered Trademark) 2000 Needle-Free Injection Management System (Biojector) for the DNA vaccine (or placebo) injection.

Subjects:

A total of 80 healthy adults will be enrolled; 40 in the 18-50 year age group and 40 in the 51-70 year age group.

Study Plan:

There are two groups in the study that are based on age. Subjects in each group will be randomized into one of two vaccination schedules. Each age group is randomized at a ratio of 1:1 to either the DNA prime-TIV boost schedule or the placebo-TIV schedule. Subjects and clinicians will be blinded to assignment to DNA vaccine or placebo for first injection until all subjects have completed Study Week 8. All subjects will receive the seasonal influenza TIV vaccine as the second injection. The initial enrollments in each group will occur no faster than 4 in the first week. Before completing enrollment, there will be a study pause with review by the Protocol Safety Review Team (PSRT) when there is at least 1 week of safety follow-up on this initial group of 8 subjects' (4 in each group) first injections. Half of the subjects will have received placebo; therefore at the time of this safety review 4 injections of the investigational DNA vaccine will have been administered. A report will be provided to the Data and Safety Monitoring Board (DSMB), which will review the study twice per year.

The protocol requires 6 clinic visits and 2 telephone follow-up contacts for all groups. This study also includes a substudy of the consent process in collaboration with the NIH Clinical Center Department of Bioethics.

Group 1 (18-50 years), 40 subjects enrolled, Group 1A: n=20 and Group 1B: n=20 will received DNA IM Biojector at Day 0 and Flulaval(Registered Trademark) IM Needle at Day 28 (plus or minus 7 days)

Group 2 (51-70 years), 40 subjects enrolled, Group 1A: n=20 and Group 2B: n=20 will received DNA IM Biojector at Day 0 and Flulaval(Registered Trademark) IM Needle at Day 28 (plus or minus 7 days)

TOTAL: 80 subjects; Day 0 injection is blinded and Day 28 is open label.

Study Duration:

Each participant will complete 24 weeks of clinical follow up.

ELIGIBILITY:
* INCLUSION CRITERIA:

A subject must meet all of the following criteria:

1. 18 to 70 years old.
2. Available for clinical follow-up through Week 24.
3. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
4. Complete an AoU prior to enrollment and verbalize understanding of all questions answered incorrectly.
5. Able and willing to complete the informed consent process.
6. Willing to donate blood for sample storage to be used for future research.
7. No evidence of previously undiagnosed clinically significant chronic diseases.
8. Physical examination and laboratory results without clinically significant findings and a Body Mass Index (BMI) greater than or equal to 18.5 and less than 40 within the 28 days prior to enrollment.

   Laboratory Criteria within 56 days prior to enrollment:
9. Hemoglobin greater than or equal to 11.5 g/dL for women; greater than or equal to 13.5 g/dL for men
10. White blood cells (WBC) = 3,300-12,000 cells/mm(3)
11. Differential either within institutional normal range or accompanied by site physician approval as a differential that is consistent with healthy volunteer status
12. Total lymphocyte count greater than or equal to 800 cells/ mm(3)
13. Platelets = 125,000 - 500,000/ mm(3)
14. Alanine aminotransferase (ALT) less than or equal to 2.5 times the upper limit of normal (ULN)
15. Serum creatinine less than or equal to 1 x ULN (less than or equal to 1.3 mg/dL for females; less than or equal to 1.4 mg/dL for males) and estimated glomerular filtration rate greater than 60.
16. Negative FDA-approved HIV blood test. [Note: Results of HIV enzyme-linked immunosorbent assay (ELISA) will be documented, but a negative HIV polymerase chain reaction (PCR) test result will be sufficient for eligibility screening of subjects with positive HIV ELISA that is due to prior participation in an HIV vaccine study].

    Female-Specific Criteria:
17. Negative human chorion gonadotropin (beta-HCG) pregnancy test (urine or serum) for women presumed to be of reproductive potential.
18. A female subject must meet one of the following criteria:

No reproductive potential because of menopause [one year without menses] or because of a hysterectomy, bilateral oophorectomy, or tubal ligation,

OR

Agrees to be heterosexually inactive at least 21 days prior to enrollment and through Week 24 of the study,

OR

Agrees to consistently practice contraception at least 21 days prior to enrollment and through Week 24 of the study by one of the following methods:

* condoms, male or female, with or without a spermicide;
* diaphragm or cervical cap with spermicide;
* intrauterine device;
* contraceptive pills, patch, implant or any other FDA-approved contraceptive method;
* male partner has previously undergone a vasectomy.

EXCLUSION CRITERIA:

A subject will be excluded if one or more of the following conditions apply.

Women Specific:

1. Breast-feeding or planning to become pregnant during the first 28 weeks after enrollment in the study.

   Subject has received any of the following substances:
2. Systemic immunosuppressive medications or cytotoxic medications, within the 12 weeks prior to enrollment. [With the exceptions that a short-acting beta-agonists in controlled asthmatics; or a short course (duration of 10 days or less or a single injection) of corticosteroids for a self-limited condition at least 2 weeks prior to enrollment in this study will not exclude study participation.]
3. Immunized with a current season FDA-approved influenza vaccine prior to enrollment.
4. Influenza infection within 6 months prior to enrollment (as assessed by clinician review of subject's self-report of a clinical course consistent with influenza).
5. Blood products within 112 days (16 weeks) prior to HIV screening
6. Immunoglobulin within 56 days (8 weeks) prior to HIV screening
7. Live attenuated vaccines within 28 days (4 weeks) prior to initial study vaccine administration
8. Investigational research agents within 28 days (4 weeks) prior to initial study vaccine administration
9. Medically indicated subunit or killed vaccines (e.g., pneumococcal, or allergy treatment with antigen injections) within 14 days (2 weeks) of initial study vaccine administration
10. Current anti-TB prophylaxis or therapy

    Subject has a history of any of the following clinically significant conditions:
11. Autoimmune disease or immunodeficiency.
12. Contraindication to receiving an FDA approved current seasonal influenza vaccination (e.g., egg allergy).
13. Serious reactions to vaccines that preclude receipt of study vaccinations as determined by the investigator.
14. Hereditary angioedema (HAE), acquired angioedema (AAE), or idiopathic forms of angioedema.
15. Asthma that is unstable or required emergent care, urgent care, hospitalization or intubation during the past two years or that requires the use of oral or intravenous corticosteroids.
16. Diabetes mellitus (type I or II), with the exception of gestational diabetes.
17. Thyroid disease that is not well controlled.
18. Idiopathic urticaria within the past 1 year.
19. Hypertension that is not well controlled by medication or is more than 145/95 at enrollment.
20. Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws.
21. Malignancy that is active or treated malignancy for which there is not reasonable assurance of sustained cure or malignancy that is likely to recur during the period of the study.
22. Seizure disorder other than: 1) febrile seizures, 2) seizures secondary to alcohol withdrawal more than 3 years ago, or 3) seizures that have not required treatment within the last 3 years.
23. Asplenia, functional asplenia or any condition resulting in the absence or removal of the spleen.
24. Guillain-Barr Syndrome.
25. Psychiatric condition that precludes compliance with the protocol; past or present psychoses; past or present bipolar disorder; disorder requiring lithium; or within 5 years prior to enrollment, a history of suicide plan or attempt.

Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2009-03-03; Primary Completion 2010-06-21 (Actual); Study Completion 2010-06-21 (Actual)

PRIMARY OUTCOMES:
safety (local and systemic reactogenicity, lab tests, AEs)

SECONDARY OUTCOMES:
lmmunogenlcity (cellular and humoral immune function assays)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Subbarao K, Murphy BR, Fauci AS. Development of effective vaccines against pandemic influenza. Immunity. 2006 Jan;24(1):5-9. doi: 10.1016/j.immuni.2005.12.005. PMID 16413916
- [Background] Luke CJ, Subbarao K. Vaccines for pandemic influenza. Emerg Infect Dis. 2006 Jan;12(1):66-72. doi: 10.3201/eid1201.051147. PMID 16494720
- [Background] Beigel JH. Influenza. Crit Care Med. 2008 Sep;36(9):2660-6. doi: 10.1097/CCM.0b013e318180b039. PMID 18679129
- [Derived] Ledgerwood JE, Hu Z, Costner P, Yamshchikov G, Enama ME, Plummer S, Hendel CS, Holman L, Larkin B, Gordon I, Bailer RT, Poretz DM, Sarwar U, Kabadi A, Koup R, Mascola JR, Graham BS; VRC 307 and VRC 309 Study Teams. Phase I clinical evaluation of seasonal influenza hemagglutinin (HA) DNA vaccine prime followed by trivalent influenza inactivated vaccine (IIV3) boost. Contemp Clin Trials. 2015 Sep;44:112-118. doi: 10.1016/j.cct.2015.08.006. Epub 2015 Aug 12. PMID 26275339
- [Derived] Enama ME, Hu Z, Gordon I, Costner P, Ledgerwood JE, Grady C; VRC 306 and 307 Consent Study Teams. Randomization to standard and concise informed consent forms: development of evidence-based consent practices. Contemp Clin Trials. 2012 Sep;33(5):895-902. doi: 10.1016/j.cct.2012.04.005. Epub 2012 Apr 20. PMID 22542645